CLINICAL TRIAL: NCT07231614
Title: Anesthetic Effectiveness of Lidocaine Versus Articaine in Dentistry. A Randomized Clinical Trial
Brief Title: Anesthetic Effectiveness of Lidocaine Versus Articaine in Dentistry
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Austral de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ArtiVsLido
Record Dates: First submitted 2025-08-27; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dental Pain
Keywords: nerve block; comparative study; exodontics; pain measurement; anesthesia infiltration
MeSH Terms: conditions — Toothache | interventions — Lidocaine; Epinephrine; Carticaine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel-group experimental study. Control group: 2% lidocaine; experimental group: 4% articaine. The RCT will be conducted in accordance with the Consolidated Standards of Reporting Trials (CONSORT 2010) guidelines.
Who Masked: Participant, Care Provider
Masking Description: Blinding will be performed by the study investigators. The RCT is a double-blind trial, where neither the operator nor the patient knows the result of the anesthesia being administered.
  The preparation of the intervention will be carried out by dividing the anesthetic cartridges, 50 for the control group (lidocaine) and 50 for the experimental group (articaine).
  Since both articaine and lidocaine are from the same manufacturer, they have the same color silicone plunger, so we will simply cover the logo with an adhesive sticker and store them in a box. To distinguish which of the tubes corresponds to articaine or lidocaine once they have the sticker, they will be assigned the same numbers that will be used to randomize each patient (1 and 2 interleaved), with No. 1 being articaine and No. 2 being lidocaine. These will be in their respective boxes with their numbering.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): Participant in this group will receive lidocaine as a local anesthetic during dental procedures.
  Interventions: Drug: lidocaine + epinephrine 1:100,000
- Articaine (Experimental): Participant in this group will receive articaine as a local anesthetic during dental procedures.
  Interventions: Drug: Articaine 4% with epinephrine 1:100,000

INTERVENTIONS:
Drug: lidocaine + epinephrine 1:100,000 — Administration of lidocaine as a local anesthetic during dental extraction.
  Arms: Lidocaine
Drug: Articaine 4% with epinephrine 1:100,000 — Administration of articaine as a local anesthetic during dental extraction.
  Arms: Articaine

SUMMARY:
Context: Lidocaine and articaine are two of the most commonly used local anesthetics in dentistry. Lidocaine has often been the anesthetic of choice in clinical practice, but in clinical experience, articaine has proven to be more effective in controlling pain during dental procedures. (Camps-Font, O. et al. 2020).

There are still unanswered questions, such as which of the two local anesthetics is more effective in reducing pain? This could lead us to discuss which one to choose to reduce costs in the dental office.

Objective: The objective of this project is to determine and compare the effectiveness of lidocaine and articaine in clinical contexts such as tooth extraction with infiltrative techniques, seeking to provide answers that will optimize the choice of anesthetic based on the patient and the procedure, thus improving pain management and reducing costs in the dental office.

Design: Randomized double-blind experimental study, parallel groups. The control group received 2% lidocaine, and the experimental group received 4% articaine. The study will be conducted in accordance with the guidelines of the Consolidated Standards of Reporting Trials (CONSORT 2010). The probabilistic sampling technique is through simple randomization. The 100 patients who meet the inclusion criteria will be randomly assigned to the control and experimental groups in a 1:1 ratio.

Expected results: articaine shows a lower percentage of extractions with anesthetic reinforcement and, therefore, a lower average number of additional tubes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical indications for simple extraction of upper and lower teeth using infiltrative anesthetic techniques.
* Patients without systemic diseases (ASA I)
* Patients with controlled systemic disease (ASA II)
* Patients with no history of hypersensitivity to anesthetics or their components (epinephrine)
* Patients with stable periodontal condition, without active infection that could affect the diffusion of the anesthetic.
* Patients with the ability to understand the procedure and provide informed consent.

Exclusion Criteria:

* Patients with uncontrolled systemic diseases ASA III and pregnant patients.
* Patients requiring trunk techniques (Gow gates, Spix, Carrea)
* Patients taking medication that affects the anesthetic response (tricyclic antidepressants, anticoagulants)
* Patients with a history of neurological or psychiatric disorders that may influence the perception of pain or anxiety.
* Patients with anatomical abnormalities in the orofacial region that interfere with the administration or action of anesthesia.
* Patients with a history of recent substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Number of tubes | immediately after the procedure
  continuous quantitative variable

SECONDARY OUTCOMES:
Pain during dislocation using the Visual Analog Scale (VAS) for pain with a minimum of 0 meaning no pain, and a maximum of 10 meaning the most severe pain ever experienced in life. | After the procedure
  Continuous quantitative variable

OTHER OUTCOMES:
Age | immediately after the procedure
  Continuous quantitative variable.
Sex | Immediately after the procedure.
  Nominal qualitative variable.

CONTACTS AND LOCATIONS:
Overall Officials: Juan E Kunstmann, Dr. Dental Surgeon Dentistry, Study Director — Universidad Austral de Chile
Locations (1):
- CESFAM Dr. Jorge Sabat, Valdivia, Los Ríos Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the trial, including demographic information, medical history relevant to the inclusion/exclusion criteria, type of anesthetic administered, and study outcome measures, will be available for secondary analyses.

REFERENCES:
- [Result] Halabi D, Escobar J, Alvarado C, Martinez N, Munoz C. Chlorhexidine for prevention of alveolar osteitis: a randomised clinical trial. J Appl Oral Sci. 2018;26:e20170245. doi: 10.1590/1678-7757-2017-0245. Epub 2018 May 7. PMID 29742264
- See also: Document that describes in detail the objectives, methodology, and procedures of the clinical trial. — https://docs.google.com/document/d/1DyLS_JgvWUSH5O9500IlCAwhV9ZJgvs4GNm3iLq89cg/edit?usp=sharing

DOCUMENTS (1):
  • Informed Consent Form (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT07231614/ICF_000.pdf